CLINICAL TRIAL: NCT06263803
Title: The Effect of Passive Music Listening in Addition to Physical Therapy on Pain, Anxiety and Quality of Life in Patients With Chronic Low Back Pain
Brief Title: The Effect of Listening to Music on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Mustafa Savaş Torlak, Asoc. Prof., KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Karataymusic
Record Dates: First submitted 2024-02-09; First posted 2024-02-16 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Masking Description: single
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): Participants in the control group will receive classical physiotherapy 5 days a week for 4 weeks (Tens 20 min, ultrasound 5 min, hotpack 20 min).
  Interventions: Other: Music listening, classic physical therapy
- Music group (Experimental): Participants in the music group will be played Pachabel Canon D major (20 minutes) and Mozart - Sonata for Two Pianos in D, K. 448 (25 minutes) during the classical physical therapy session, free from external sounds (max 70 dB through headphones).
  Interventions: Other: Music listening, classic physical therapy

INTERVENTIONS:
Other: Music listening, classic physical therapy — Participants will listen to the music pieces Pachabel Canon in D major (20 minutes) and Mozart - Sonata for Two Pianos in D, K. 448 (25 minutes), free from external sounds (max 70 dB through headphones).

SUMMARY:
The effects of passive music listening on pain, anxiety and quality of life in patients with chronic low back pain in addition to physical therapy will be examined.

DETAILED DESCRIPTION:
The aim of the study was to investigate the effects of passive music listening in addition to physical therapy on pain, anxiety and quality of life in patients with chronic low back pain.There is no study in the literature examining the relationship between music listening and physical therapy in chronic back pain. Since our study will be the first to investigate the subject, we foresee that it is scientifically important and will shed light on future studies. In addition, national or international publications are planned after the study is completed.

ELIGIBILITY:
Inclusion Criteria:

patients with LBP for more than 3 months with pain severity of 5 or greater according to the visual analogue scale (VAS)

Exclusion Criteria:

individuals who regularly take painkillers or anti-depressant and cortisone; pregnant individuals; and individuals having severe chronic illness and spine surgery were excluded from the study

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Beck anxiety inventory | baseline and 4 weeks
  The Beck Anxiety Inventory (BAI) consists of 21 self-reported items (four-point scale) used to assess the intensity of physical and cognitive anxiety symptoms during the past week. Scores may range from 0 to 63: minimal anxiety levels (0-7), mild anxiety (8-15), moderate anxiety (16-25), and severe anxiety (26-63).
Visual Analogue Scale | baseline and 4 weeks
  A Visual Analogue Scale (VAS) is one of the pain rating scales used for the first time in 1921 by Hayes and Patterson. It is often used in epidemiologic and clinical research to measure the intensity or frequency of various symptoms. For example, the amount of pain that a patient feels ranges across a continuum from none to an extreme amount of pain.
Short From-36 | baseline and 4 weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study for the objective measure of the quality of life.
  It comprises 36 questions that cover eight domains of health:
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions

CONTACTS AND LOCATIONS:
Locations (1):
- Mustafa Savaş Torlak, Karatay, Eyalet/Yerleşke, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided